CLINICAL TRIAL: NCT06531759
Title: Efficacy of Fentanyl Soaked Nasal Packs on Postoperative Pain in Nasal Surgeries.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Mahmoud Abd ElMonem Mahmoud, Aya Mahmoud Abd ElMonem, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pain after nasal surgeries
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients undergoing nasal surgeries requiring bilateral nasal packs. (Other): After performing the required nasal surgery, hydroxylated polyvinyl acetate packs (known as merocele packs) will be applied bilaterally in patients. The merocele on the left side will be injected with 5 ml volume of normal saline, while The merocele pack in the right side will be injected with 5 ml volume of the diluted fentanyl solution (1ml of fentanyl 50mcg diluted in 10 ml of normal saline).
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Fentanyl soaked nasal packs.

SUMMARY:
Efficacy of fentanyl soaked nasal packs on postoperative pain in nasal surgeries.

DETAILED DESCRIPTION:
Postoperative pain is one of the commonest feared surgical side effect which can lead to patient dissatisfaction. It occurs due to a combination of inflammatory reaction and an injury to neural tissue caused by the surgical incision. Anterior nasal packing is not an innocuous procedure. It causes discomfort/pain (especially upon removal), nasal mucosa trauma, epiphora, local infection, discomfort in swallowing, sleep disturbances and, very rarely, toxic shock and vagal reflex. Although systemic opioids are traditionally used in the management of postoperative pain, their use is still limited by their possible side effects. Opioid drugs mimic the actions of the endogenous opioid peptides by interacting with specific receptors, the opioid receptors which are μ, δ and κ. The μ receptor is important in sensory processing, including the modulation of nociceptive stimuli, extrapyramidal functioning and in limbic and neuroendrocine regulation. There are two subtypes of the μ receptor, a high-affinity μ receptor and a low-affinity μ2 receptor. Recently a third μ subtype has been described that binds opioid alkaloids such as morphine, but has essentially no, or exceedingly low, affinity for the naturally occurring endogenous opioid peptides or non-alkaloid opioids such as fentanyl. Based on the hypothesis that mu (μ) opioid receptor expression increases at the site of inflammation. our study aims to assess the analgesic effect produced by local application of fentanyl through fentanyl soaked nasal packs following different nasal surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing nasal surgeries requiring bilateral nasal packs.
2. Patients 18 years or older.

Exclusion Criteria:

1. Patients in whom fentany is contraindicated such as respiratory comorbidites (COPD and Asthma), hypersensitivity to fentanyl, liver diseases or had previous biliary tract surgeries
2. Systemic medical problems interfering with surgery.
3. Patients with traumatic conditions e.g fracture face or fracture nasal bone.
4. patients who refuse to take part in the study.
5. Patients with different nasal pathology in both sides e.g if partial turbinectomy is indicated in one side of the nose or patients with unilateral nasal polyp.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy of fentanyl soaked nasal packs on postoperative pain in nasal surgeries | 24 hours postoperatively
  Assessment of pain intensity will be done using The 11-point Numeric pain rating scale, subjects will be asked to give a pain score ranging from 0 to 10 interpreted as 0 is no pain and 10 is the worst pain they ever felt at intervals of 3, 6, 12 and 24 hours postoperatively.